CLINICAL TRIAL: NCT03449576
Title: Efficacy and Neural Mediators of Response to Trauma Management Therapy for PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: D2354-R
Record Dates: First submitted 2018-02-15; First posted 2018-02-28 (Actual); Results first posted 2024-07-01 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-03

CONDITIONS: PTSD
Keywords: PTSD; neuroimaging; fMRI; veterans; exposure therapy; treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Implosive Therapy; Psychotherapy, Group

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trauma Management Therapy (Experimental): Trauma Management Therapy (TMT) consists of a combination of 12 sessions of individualized exposure therapy and 24 sessions of group-based social and emotion rehabilitation.
  Interventions: Other: Trauma Management Therapy
- Exposure Therapy with Psychoeducation (Active Comparator): Exposure Therapy with Psychoeducation (EXP+EDU) consists of a combination of 12 sessions of individualized exposure therapy and 24 session of group-based psychoeducation.
  Interventions: Other: Exposure Therapy with Psychotherapy group

INTERVENTIONS:
Other: Trauma Management Therapy — Trauma Management Therapy (TMT) consists of a combination of 12 sessions of individualized exposure therapy and 24 sessions of group-based social and emotion rehabilitation.
  Other Names: TMT
  Arms: Trauma Management Therapy
Other: Exposure Therapy with Psychotherapy group — Exposure Therapy with Psychoeducation (EXP+EDU) consists of a combination of 12 sessions of individualized exposure therapy and 24 session of group-based psychoeducation.
  Other Names: EXP+GRP
  Arms: Exposure Therapy with Psychoeducation

SUMMARY:
Social difficulties are serious and frequent complicating factors in the treatment of post-traumatic stress disorder (PTSD). To better understand how treatment of post-traumatic stress disorder impacts neural mechanisms of social cognition, the investigators are examining behavior and brain processes associated with response to Trauma Management Therapy. Understanding the behavioral and neural impact of psychotherapy may contribute to development of more effective treatments for PTSD.

DETAILED DESCRIPTION:
PTSD is associated with significant interpersonal difficulties that interfere with functioning. As such, this work is intended to evaluate the empirical support for a novel treatment that fills a significant gap in the treatment options available to Veterans with PTSD who suffer with interpersonal difficulties. In this study the investigators will (i) evaluate the efficacy of Trauma Management Therapy (TMT) for treating PTSD-related interpersonal dysfunction, as well as PTSD-related fear and anxiety, and (ii) evaluate neural mediators of clinical improvements associated with TMT.

This work will provide insights into the mechanisms by which treatments may lead to improvements in social functioning, informing both the biological basis of psychotherapy and the development and refinement of alternative therapeutic interventions targeting social impairments.

Treatment seeking Veterans with PTSD will be randomized to one of two treatments: (i) Trauma Management Therapy, consisting of 12 sessions of individualized exposure therapy followed by 24 sessions of group-based social and emotional rehabilitation, or (ii) Exposure + Comparison Treatment Group consisting of 12 sessions of individualized exposure therapy followed by 24 sessions of group-based psychotherapy. Veterans enrolled in both the TMT and EXP+GRP arms will undergo functional neuroimaging as they engage in an emotional image viewing task, as well as two social interaction tasks. Neurobehavioral assessments will be made prior to and following completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female veterans of all ethnicities
* Meet diagnostic criteria for post-traumatic stress disorder (assessed by study staff)
* Fluent in English
* Able to see computer display clearly
* Able to provide informed consent
* Able to follow written or verbal instructions

Exclusion Criteria:

* history of seizures
* history of stroke
* Cushing's syndrome
* history of moderate to severe traumatic brain injury
* electroconvulsive therapy within 5 years
* history of chemotherapy for cancer
* contraindications to fMRI
* pregnancy
* diagnosis of schizophrenia, schizoaffective disorder, delusional disorder and/or organic psychosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brooks King-Casas, PhD, Principal Investigator — Salem VA Medical Center, Salem, VA
Locations (1):
- Salem VA Medical Center, Salem, VA, Salem, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trauma Management Therapy | Exposure Therapy With Psychoeducation
Started | 40 | 29
Completed | 29 | 24
Not Completed | 11 | 5

BASELINE CHARACTERISTICS:
Population: Treatment seeking Veterans with Post-Traumatic Stress Disorder (PTSD) assigned to each treatment group
Groups:
- Total: Total of all reporting groups
Arm/Group | Trauma Management Therapy | Exposure Therapy With Psychoeducation | Total
Number analyzed (Participants) | 40 | 29 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.65 (9.40) | 43.83 (10.35) | 48.36 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 28 | 21 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 38 | 26 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 17 | 8 | 25
  White | 19 | 19 | 38
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician-Administered PTSD Scale for DSM-5
Description: The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5; Weathers et al. 2013; 2017) is a 20 item semi-structured instrument for the diagnosis and assessment of severity of posttraumatic stress disorder (PTSD). Each DSM-5 item is rated on a 0 (absent) to 4 (extreme/incapacitating) scale, and total score is calculated by summing severity scores across items. Total CAPS-5 severity can range from 0 to 80. [edited 2/24/24: Higher scores mean a worse outcome.]
Time Frame: CAPS-5 will be assessed at two time-points per participant: before starting treatment i.e. pre-treatment (week 0) and at completion of treatment, i.e. post-treatment (week 8).
Population: Data analysis at pre-treatment was limited to participants who had completed this measure. At post-treatment, analysis was limited to participants who had begun treatment and had completed this measure.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Trauma Management Therapy | Exposure Therapy With Psychoeducation
Number analyzed (Participants) | 29 | 24
score on a scale
  Pre-treatment: number analyzed (Participants) | 18 | 24
  Pre-treatment | 38.39 (2.834358) | 35.67 (1.76075)
  Post-treatment: number analyzed (Participants) | 13 | 12
  Post-treatment | 27.15 (4.324715) | 29.31 (2.813394)
Statistical Analysis 1: Comparison: Trauma Management Therapy vs Exposure Therapy With Psychoeducation; Test of prediction of dependent variable -- the CAPS score-- with the interaction between Visit (pre/post) and treatment type (TMT vs. EXP+EDU), as well as independent variable, age; Test type: Superiority; p = 0.4154, Regression, Linear — This P value is the interaction term between Visit and Treatment; Slope = 5.3846, Standard Error of Mean 6.5525 — This is the beta value for the interaction term between Visit and Treatment

2. Primary Outcome: Change in Social Adjustment Scale - Self-Report
Description: The Social Adjustment Scale (SAS; Weissman & Bothwell, 1976) is a 54 item self-report measure that assesses social adjustment in six social areas of functioning including work, social and leisure activities, extended family, marital, parental, and family. Each item is rated on a five point scale, and within each of domain items are averaged. Thus, scores in each domain can range between 1 (high social adjustment) and 5 (low social adjustment). [edited 2/24/24 Higher scores mean a worse outcome.]
Time Frame: SAS will be assessed at two time-points: before starting treatment i.e. pre-treatment (week 0) and at completion of treatment, i.e. post-treatment (week 8).
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mean score on a scale
Arm/Group | Trauma Management Therapy | Exposure Therapy With Psychoeducation
Number analyzed (Participants) | 29 | 24
mean score on a scale
  Pre-treatment: number analyzed (Participants) | 29 | 23
  Pre-treatment | 2.855 (0.1321421) | 3.168 (0.1061295)
  Post-treatment: number analyzed (Participants) | 24 | 9
  Post-treatment | 2.953 (0.1869682) | 3.289 (0.125691)
Statistical Analysis 1: Comparison: Trauma Management Therapy vs Exposure Therapy With Psychoeducation; Test of prediction of dependent variable -- the SAS-SR score-- with the interaction between Visit (pre/post) and Treatment type (TMT vs. EXP+EDU), as well as independent variable, age; Test type: Superiority; p = 0.4636, Regression, Linear — This P value is the interaction term between Visit and Treatment; Slope = 0.267397, Standard Error of Mean 0.362521 — This is the beta value for the interaction term between Visit and Treatment

3. Primary Outcome: Change in PTSD Checklist for DSM-5
Description: The PTSD Checklist for DSM-5 (PCL-5; Weathers et al., 2013; Bovin et al., 2016) is a 20 item self-report measure assessing DSM-5 PTSD symptom severity. Each DSM-5 item is rated on a 0 (absent) to 4 (extreme/incapacitating) scale, and total score is calculated by summing severity scores across items. Total CAPS-5 severity can range from 0 to 80. Higher scores mean a worse outcome.
Time Frame: The PCL-5 will be assessed at two time-points: before starting treatment i.e. pre-treatment (week 0) and at completion of treatment, i.e. post-treatment (week 8).
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Trauma Management Therapy | Exposure Therapy With Psychoeducation
Number analyzed (Participants) | 29 | 24
score on a scale
  Pre-treatment | 53.66 (2.594175) | 56.92 (2.917909)
  Post-treatment: number analyzed (Participants) | 24 | 17
  Post-treatment | 40.04 (3.610813) | 46.53 (4.15784)
Statistical Analysis 1: Comparison: Trauma Management Therapy vs Exposure Therapy With Psychoeducation; Test of prediction of dependent variable -- the PCL score-- with the interaction between Visit (pre/post) and treatment type (TMT vs. EXP+EDU), as well as independent variable, age; Test type: Superiority; p = 0.735129, Regression, Linear — This P value is the interaction term between Visit and Treatment; Slope = 2.3355, Standard Error of Mean 6.8791 — This is the beta value for the interaction term between Visit and Treatment

4. Secondary Outcome: Change in Aggression Questionnaire
Description: Change in Aggression Questionnaire (AQ; Buss & Warren, 2000) is a 34 item self-report measure that assesses severity of self-perceived aggression and anger. Each item is rated on a 1 (Not at all like me) to 5 (Completely like me) scale, and scores of all items are summed. Scores can range from 34 to 170. Higher scores mean a worse outcome.
Time Frame: AQ will be assessed at two time-points: before starting treatment i.e. pre-treatment (week 0) and at completion of treatment, i.e. post-treatment (week 8).
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Trauma Management Therapy | Exposure Therapy With Psychoeducation
Number analyzed (Participants) | 29 | 24
score on a scale
  Pre-treatment | 59 (1.83896) | 64.62 (1.715036)
  Post-treatment: number analyzed (Participants) | 24 | 17
  Post-treatment | 58.92 (2.066746) | 62.18 (3.193785)
Statistical Analysis 1: Comparison: Trauma Management Therapy vs Exposure Therapy With Psychoeducation; Test of prediction of dependent variable -- the AQ score-- with the interaction between Visit (pre/post) and treatment type (TMT vs. EXP+EDU), as well as independent variable, age; Test type: Superiority; p = 0.580, Regression, Linear — This P value is the interaction term between Visit and Treatment; Slope = -2.64908, Standard Error of Mean 4.76601 — This is the beta value for the interaction term between Visit and Treatment

5. Secondary Outcome: Change in Interpersonal Trust Scale
Description: Change in Interpersonal Trust Scale (ITS; Rotter, 1967) is a 25 item self-report measure that assesses trust within relationships. Each item is rated on a 1 (low trust) to 5 (high trust) scale, and total scores can range from 25 to 125. [edited 2/24/24: Higher scores mean a better outcome.]
Time Frame: ITS will be assessed at two time-points: before starting treatment i.e. pre-treatment (week 0) and at completion of treatment, i.e. post-treatment (week 8).
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Trauma Management Therapy | Exposure Therapy With Psychoeducation
Number analyzed (Participants) | 29 | 24
score on a scale
  Pre-treatment | 60.21 (2.266907) | 57.54 (1.917671)
  Post-treatment: number analyzed (Participants) | 24 | 17
  Post-treatment | 63.33 (2.491774) | 60.41 (4.027533)
Statistical Analysis 1: Comparison: Trauma Management Therapy vs Exposure Therapy With Psychoeducation; Test of prediction of dependent variable -- the ITS score-- with the interaction between Visit (pre/post) and treatment type (TMT vs. EXP+EDU), as well as independent variable, age; Test type: Superiority; p = 0.808, Regression, Linear — This P value is the interaction term between Visit and Treatment; Slope = 1.3946, Standard Error of Mean 5.7193 — This is the beta value for the interaction term between Visit and Treatment

ADVERSE EVENTS:
Time Frame: 7 months, 3 weeks
Description: Participants were assessed across a period of seven months and three weeks, including seven weeks of treatment and a six month follow-up period.
Arm/Group | Trauma Management Therapy | Exposure Therapy With Psychoeducation
All-Cause Mortality (participants affected / at risk) | 2/40 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/40 | 1/29
Other Adverse Events (participants affected / at risk) | 0/40 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trauma Management Therapy (N=40) | Exposure Therapy With Psychoeducation (N=29)
Syncopal episode (Cardiac disorders) | 0 | 1
Psychiatric hospitalization (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT03449576/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT03449576/SAP_001.pdf
  • Informed Consent Form (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/76/NCT03449576/ICF_002.pdf